CLINICAL TRIAL: NCT00603343
Title: Treatment With Propiverine in Children Suffering From Non-Neurogenic Overactive Bladder and Urinary Incontinence: Results of a Randomized Placebo-Controlled Phase III Clinical Trial
Brief Title: Propiverine in Children Suffering From Non-Neurogenic Overactive Bladder and Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: APOGEPHA Arzneimittel GmbH (Industry)
Responsible Party: APOGEPHA, APOGEPHA Arzneimittel GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT-Number 200400124330
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2008-01

CONDITIONS: Overactive Bladder; Urinary Incontinence; Children
Keywords: antimuscarinics; children; overactive bladder; propiverine; urinary incontinence; urotherapy
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — propiverine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Mictonetten 5 mg, coated tablet
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mictonetten 5 mg, coated tablet — propiverine 10 mg b.i.d. (17-27.9 kg BW) or propiverine 15 mg b.i.d. (28-45.0 kg BW)
  Other Names: Mictonetten
  Arms: 1
Drug: placebo — placebo corresponding to body weight
  Arms: 2

SUMMARY:
The study was conducted between 2004 and 2006 to prove efficacy and tolerability of the antimuscarinic propiverine compared to placebo in children suffering from non-neurogenic overactive bladder and urinary incontinence.

DETAILED DESCRIPTION:
This clinical trial showed superior efficacy of propiverine over placebo and convincing tolerability for the treatment of children suffering from OAB and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* voiding frequency 8 or above per day
* at least one incontinence episode per day
* age between 5-10 years
* body weight between 17 and 45 kg

Exclusion Criteria:

* normal age expected bladder capacity
* PVR more than 10 ml
* dysfunctional voiding
* neurogenic disorders
* UTI, constipation

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2004-06; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
voiding frequency | before therapy and at end of therapy

SECONDARY OUTCOMES:
voided volume | before and at end of treatment
incontinence episodes per day | before and at end of therapy
safety parameters: acute urinary retention, post void residual urine, urinalysis, ECG, blood pressure, pulse rate | before and at end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Marschall-Kehrel, MD, Principal Investigator — urologist

REFERENCES:
- [Derived] Marschall-Kehrel D, Feustel C, Persson de Geeter C, Stehr M, Radmayr C, Sillen U, Strugala G. Treatment with propiverine in children suffering from nonneurogenic overactive bladder and urinary incontinence: results of a randomized placebo-controlled phase 3 clinical trial. Eur Urol. 2009 Mar;55(3):729-36. doi: 10.1016/j.eururo.2008.04.062. Epub 2008 May 7. PMID 18502028